CLINICAL TRIAL: NCT03749252
Title: Pharmacokinetics, Safety and Efficacy of a New Gadolinium-based Contrast Agent, P03277, in Pediatric Patients From 2 to 17 Years of Age Undergoing Central Nervous System Contrast-enhanced MRI
Brief Title: Pharmacokinetics, Safety and Efficacy of P03277 in Pediatric Patients Undergoing Central Nervous System Contrast-enhanced MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GDX-44-007; 2018-001516-30 (EudraCT Number)
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Central Nervous System Indication; Pediatric Patients; Body Indication
MeSH Terms: interventions — gadopiclenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CNS Cohort 2-6 years (Experimental): Pediatric patients aged 2-6 years undergoing CNS contrast-enhanced MRI
  Interventions: Drug: P03277
- CNS Cohort 7-11 years (Experimental): Pediatric patients aged 7-11 years undergoing CNS contrast-enhanced MRI
  Interventions: Drug: P03277
- CNS Cohort 12-17 years (Experimental): Pediatric patients aged 12-17 years undergoing CNS contrast-enhanced MRI
  Interventions: Drug: P03277
- Body Cohort 2-6 years (Experimental): Pediatric patients aged 2-6 years undergoing contrast-enhanced MRI of other body organs (head and neck, thorax, abdomen, pelvis or musculoskeletal system)
  Interventions: Drug: P03277
- Body Cohort 7-11 years (Experimental): Pediatric patients aged 7-11 years undergoing contrast-enhanced MRI of other body organs (head and neck, thorax, abdomen, pelvis or musculoskeletal system)
  Interventions: Drug: P03277
- Body Cohort 12-17 years (Experimental): Pediatric patients aged 12-17 years undergoing contrast-enhanced MRI of other body organs (head and neck, thorax, abdomen, pelvis or musculoskeletal system)
  Interventions: Drug: P03277

INTERVENTIONS:
Drug: P03277 — A dose of 0.05 mmol/kg body weight (0.1 mL/kg body weight) of P03277 will be administered to each patient in a single intravenous injection.
  Other Names: gadopiclenol

SUMMARY:
This is a pharmacokinetics (PK), open-label, uncontrolled, multicenter phase II trial with age-staggered approach.

The primary objective is to evaluate the PK profile of gadopiclenol in plasma following single IV injection of 0.05 mmol/kg body weight (BW) in pediatric population aged from 2 to 17 years undergoing CNS contrast-enhanced MRI (CNS cohort).

DETAILED DESCRIPTION:
A population PK approach and an age-down staggered approach will be used. Patients will be recruited into 3 predefined age groups: 12-17, 7-11 and 2-6 years. The inclusions will start with the older group (Adolescents, 12-17 years), followed by Preadolescents (7-11 years) and finally Young Children (2-6 years of age).

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, the patient had to meet all the following criteria:

1. Female or male pediatric patient aged 2 to 17 years,
2. Patient with known or suspected lesion(s) scheduled to undergo routine contrast-enhanced MRI of CNS or of other organs including at least one organ among head and neck, thorax, abdomen, pelvis or musculoskeletal system (including extremities),
3. Patient whose parent(s) or legal guardian having read the information, provided their consent to patient's participation in writing by dating and signing the informed consent prior to any trial related procedure being conducted,
4. Patient with capacity of understanding who received age- and maturity-appropriate information and provided his/her assent to participate in the trial (as required by national regulations),
5. Patient affiliated to national health insurance according to local regulatory requirements.

Non-inclusion Criteria:

Patients could not be included in the study if they presented with one or more of the following non-inclusion criteria:

1. Patient planned for treatment or procedure (e.g., surgery) that would prevent obtaining the required blood samples or performing other trial procedures between the screening visit and up to 1 day after gadopiclenol administration,
2. Patient undergoing treatment or procedure (e.g., diuretics, clinically significant blood loss or blood transfusion) preceding or subsequent to gadopiclenol administration that would alter gadopiclenol PK parameters,
3. Patient with acute or chronic renal insufficiency defined as estimated Glomerular Filtration Rate (eGFR) out of age-adjusted normal ranges (eGFR calculated with bedside Schwartz equation),
4. Patients referred for MR Angiography,
5. Patient with history of bleeding disorder,
6. Patient with known severe liver disease,
7. Patient with known cardiac disease (e.g., heart rhythm anomalies, long QT syndrome),
8. Patient with any clinically significant abnormal 12-lead ECG that in the Investigator's opinion would affect the safety evaluation or place the patient at risk,
9. Patient with electrolyte or fluid imbalance that at Investigator's judgment presents undue risk assessed within 1 month prior to gadopiclenol administration,
10. Patient undergoing a change in chemotherapy within 1 day prior to or 1 day after gadopiclenol administration,
11. Patient who received any other contrast agent for CT and/or MRI within 1 week prior to or 1 week after gadopiclenol administration,
12. Patient with contraindication for MRI such as iron metal implants (e.g., aneurysm clips, pacemaker),
13. Patient with history of anaphylactoid or anaphylactic reaction to any allergen including drugs,
14. Patient with history of hypersensitivity caused by any contrast media / agents (iodinated or gadolinium-based),
15. Patient with known contraindication(s) to the use of any GBCA,
16. Pregnant or breast-feeding female patient (female patient with childbearing potential [who experienced menarche] must have a negative urine pregnancy test within 24 hours prior to gadopiclenol administration and must be using medically approved contraception* if sexually active),
17. Patient with anticipated, current or past condition (medical, psychological, social or geographical) that would compromise the patient's safety or her/his ability to participate to the whole trial,
18. Patient unlikely to comply with the protocol, e.g., uncooperative attitude of parent(s) or legal guardian, inability to return for follow-up visits and unlikelihood of completing the trial,
19. Having participated in a clinical trial and having received any investigational product within 7 days prior to gadopiclenol administration or planned during the trial,
20. Patient previously included in this trial,
21. Patient related to the Investigator or any other trial staff or relative directly involved in the trial conduct.

    * medically approved contraception methods include: female sterilization, use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception, placement of an Intrauterine Device (IUD) or Intrauterine System (IUS), barrier methods of contraception (condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elżbieta Jurkiewicz, MD, Principal Investigator — Instytut Pomnik
Locations (16):
- Bulgaria (3):
  - MHAT Central Onco Hospital Ltd, Plovdiv
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - MHAT Dr. Stoyan Kirkovich, Stara Zagora
- Hungary (3):
  - Semmelweis Egyetem II. sz Gyermekgyogyaszati Klinika, Budapest
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - B.-A.-Z. Megyei Korhaz Gyermek-Egeszsegugyi Kozpont, Miskolc
- Poland (6):
  - Szpital Uniwersytecki nr 1 w Bydgoszczy im. dr Jurasza, Oddział Kliniczny Chirurgii Ogólnej i Onkologicznej Dzieci i Młodzieży, Bydgoszcz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Uniwersytecki Szpital Dziecięcy w Lublinie, Lublin
  - Klinika Chirurgii Dziecięcej, Rzeszów
  - Instytut "Pomnik -Centrum Zdrowia Dziecka", Warsaw
  - Zakład Radiologii PediatrycznejSamodzielny Publ. Dziecięcy Szp. Kliniczny w Warszawie, Warsaw
- Slovakia (3):
  - II. Detská klinika SZU, Detská fakultná nemocnica s poliklinikou Banská Bystrica, Banská Bystrica
  - Klinika detí a dorastu JLF UK a UNM, Univerzitná nemocnica Martin, Martin
  - Faculty hospital Nitra, Clinic of neonates, children and adolescents, Nitra
- Children's City Clinical Hospital, Dnipro, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jurkiewicz E, Tsvetkova S, Grinberg A, Pasquiers B. Pharmacokinetics, Safety, and Efficacy of Gadopiclenol in Pediatric Patients Aged 2 to 17 Years. Invest Radiol. 2022 Aug 1;57(8):510-516. doi: 10.1097/RLI.0000000000000865. Epub 2022 Mar 2. PMID 35318970

RESULTS

PARTICIPANT FLOW:
Groups:
- CNS & Body Cohorts 2-6 Years: Pediatric patients aged 2-6 years undergoing CNS or Body contrast-enhanced MRI
  P03277: A dose of 0.05 mmol/kg body weight (0.1 mL/kg body weight) of P03277 will be administered to each patient in a single intravenous injection.
- CNS & Body Cohorts 7-11 Years: Pediatric patients aged 7-11 years undergoing CNS or Body contrast-enhanced MRI
  P03277: A dose of 0.05 mmol/kg body weight (0.1 mL/kg body weight) of P03277 will be administered to each patient in a single intravenous injection.
- CNS & Body Cohorts 12-17 Years: Pediatric patients aged 12-17 years undergoing CNS or Body contrast-enhanced MRI
  P03277: A dose of 0.05 mmol/kg body weight (0.1 mL/kg body weight) of P03277 will be administered to each patient in a single intravenous injection.
Period: Overall Study
Arm/Group | CNS & Body Cohorts 2-6 Years | CNS & Body Cohorts 7-11 Years | CNS & Body Cohorts 12-17 Years
Started | 26 | 23 | 31
Completed | 26 | 23 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received gadopiclenol administration and underwent CNS or Body MRI
Groups:
- Total: Total of all reporting groups
Arm/Group | CNS & Body Cohorts 2-6 Years | CNS & Body Cohorts 7-11 Years | CNS & Body Cohorts 12-17 Years | Total
Number analyzed (Participants) | 26 | 23 | 31 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (1.3) | 8.8 (1.2) | 14.3 (1.6) | 9.3 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 19 | 39
  Male | 19 | 10 | 12 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 23 | 31 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 26 | 23 | 31 | 80
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Elimination Half-life
Description: P03277 pharmacokinetic parameters in plasma were determined from the population PK model.
  This outcome was assessed only for the CNS cohort.
Time Frame: 4 blood samples per patient were taken post-injection for PK analysis, one within each window: 1 min to 20 min, 30 min to 45 min, 2 to 3 hours and 7 to 8 hours
Population: All patients of the CNS cohort who received gadopiclenol administration except one patient, whose PK blood samples were assessed out of stability period
Measure: Median (Full Range); unit: hours
Arm/Group | CNS Cohort 2-6 Years | CNS Cohort 7-11 Years | CNS Cohort 12-17 Years
Number analyzed (Participants) | 20 | 20 | 19
hours | 1.29 [0.69 to 3.38] | 1.48 [0.83 to 3.20] | 1.77 [1.00 to 3.57]

2. Primary Outcome: Total Clearance
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: L/h/kg
Arm/Group | CNS Cohort 2-6 Years | CNS Cohort 7-11 Years | CNS Cohort 12-17 Years
Number analyzed (Participants) | 20 | 20 | 19
L/h/kg | 0.12 [0.05 to 0.28] | 0.10 [0.04 to 0.24] | 0.08 [0.04 to 0.20]

3. Primary Outcome: Central Volume of Distribution
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: L/kg
Arm/Group | CNS Cohort 2-6 Years | CNS Cohort 7-11 Years | CNS Cohort 12-17 Years
Number analyzed (Participants) | 20 | 20 | 19
L/kg | 0.12 [0.06 to 0.26] | 0.12 [0.06 to 0.24] | 0.11 [0.05 to 0.24]

4. Primary Outcome: Peripheral Volume of Distribution
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: L/kg
Arm/Group | CNS Cohort 2-6 Years | CNS Cohort 7-11 Years | CNS Cohort 12-17 Years
Number analyzed (Participants) | 20 | 20 | 19
L/kg | 0.06 [0.06 to 0.06] | 0.06 [0.06 to 0.06] | 0.06 [0.06 to 0.06]

5. Primary Outcome: Area Under the Curve
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg.h/L
Arm/Group | CNS Cohort 2-6 Years | CNS Cohort 7-11 Years | CNS Cohort 12-17 Years
Number analyzed (Participants) | 20 | 20 | 19
mg.h/L | 403.16 (93.35) | 477.25 (105.71) | 582.30 (122.08)

6. Primary Outcome: Simulated Concentrations 10 Minutes Post-injection
Description: as for outcome 1
Time Frame: 10 minutes post-injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CNS Cohort 2-6 Years | CNS Cohort 7-11 Years | CNS Cohort 12-17 Years
Number analyzed (Participants) | 20 | 20 | 19
mg/L | 302.11 (44.68) | 327.20 (47.95) | 349.15 (52.59)

7. Primary Outcome: Simulated Concentrations 20 Minutes Post-injection
Description: as for outcome 1
Time Frame: 20 minutes post-injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CNS Cohort 2-6 Years | CNS Cohort 7-11 Years | CNS Cohort 12-17 Years
Number analyzed (Participants) | 20 | 20 | 19
mg/L | 234.88 (30.18) | 259.67 (32.02) | 285.16 (35.35)

8. Primary Outcome: Simulated Concentrations 30 Minutes Post-injection
Description: as for outcome 1
Time Frame: 30 minutes post-injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CNS Cohort 2-6 Years | CNS Cohort 7-11 Years | CNS Cohort 12-17 Years
Number analyzed (Participants) | 20 | 20 | 19
mg/L | 188.26 (25.10) | 211.20 (25.82) | 237.25 (26.97)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from informed consent signature untill the end of the study (up to 120 days after gadopiclenol administration).
Description: The Safety Set included all patients who had received at least one injection of gadopiclenol.
Arm/Group | CNS & Body Cohorts 2-6 Years | CNS & Body Cohorts 7-11 Years | CNS & Body Cohorts 12-17 Years
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/23 | 2/31
Other Adverse Events (participants affected / at risk) | 4/26 | 6/23 | 4/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNS & Body Cohorts 2-6 Years (N=26) | CNS & Body Cohorts 7-11 Years (N=23) | CNS & Body Cohorts 12-17 Years (N=31)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNS & Body Cohorts 2-6 Years (N=26) | CNS & Body Cohorts 7-11 Years (N=23) | CNS & Body Cohorts 12-17 Years (N=31)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 1 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Long QT syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Procedural Anxiety (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT03749252/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03749252/SAP_001.pdf